CLINICAL TRIAL: NCT02282709
Title: Effect of ASV and DCV Therapy on the Quality of Immune Status in Chronic HCV Patients
Acronym: ImmunoDual
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Foundation_LiverR
Record Dates: First submitted 2014-10-23; First posted 2014-11-04 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Hepatitis C
Keywords: Immunity
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — daclatasvir; asunaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daclatasvir and asunaprevir (Experimental): daclatasvir 60 mg once daily asunaprevir 100 mg BID
  Interventions: Drug: Daclatasvir; Drug: asunaprevir

INTERVENTIONS:
Drug: Daclatasvir — 60 mg once daily
Drug: asunaprevir — 100 mg BID

SUMMARY:
Rationale: Chronic HCV infection is characterised by a weak HCV specific CD8+ T cell response, due to continuous pressure of high viral load. Treatment of chronic HCV patients with ASV and DCV will result in a significant drop in HCV viral load. At present, no information is available on the immunological effects of treatment with ASV and DCV, nor on the early effects of viral load reduction caused by a compound that is thought not to possess direct immunomodulatory effects. This information will be crucial for a better understanding of the mechanisms that may limit the effectiveness of treatment, occurrence of viral rebound or relapses during, at the end of treatment or during the follow up period.

Objective: To evaluate in detail the functionality of immune cells in blood in chronic HCV patients before, during and after treatment with ASV and DCV, in an IFN-free regimen.

Study design: This is an investigator-initiated single center open label study with one arm of 12 patients.

Study population: Adult chronic HCV patients with genotype 1b, who are previous non-responders to the treatment.

Intervention (if applicable): All patients will be treated with twice daily a 200 mg oASV and once daily a 60 mg DCV for 24 weeks.

Main study parameters/endpoints:

1. Phenotype and function of blood leukocytes during treatment; frequency of HCV-specific T cells, NK cells and monocytes
2. Gene expression levels of leukocyte populations before, during and after treatment
3. Gene expression levels of the type I IFN signaling pathway on whole blood samples
4. Serum cytokines levels using multiplex platforms

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age, with a chronic hepatitis C - genotype 1b infection
* Patients are non-responders to previous treatment with peginterferon or conventional interferon plus ribavirin combination therapy
* High viral load (>400,000 IU/ml)
* Indication for antiviral therapy of hepatitis C according to current clinical guidelines
* Written informed consent

Exclusion Criteria:

* Decompensated cirrhosis (Child-Pugh Grade B or C)
* Hepatic imaging (ultrasound, CT or MRI) with the evidence of hepatocellular carcinoma within the last 3 months.
* Females who are pregnant or breast-feeding
* History or other evidence of severe illness, malignancy or any other condition which would make the patient, in the opinion of the investigators, unsuitable for the study
* Co-infections with human immunodeficiency virus (HIV) or Hepatitis B virus (HBV)
* Presence of contra-indications for antiviral therapy with ASV and DCV:
* Interfering substance abuse, such as high alcohol intake (indicator: 28 drinks/ week)
* Any exposure to NS3 protease inhibitors or NS5A polymerase inhibitors
* Treatment with peginterferon/ ribavirin within 6 months before start of therapy
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating and completing in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
HCV-specific T cell phenotype and function (a composite measure of (I) HCV-specific T-cell frequency and (II) phenotypic expression of memory markers and (III) inhibitory receptor markers | 1 year
NK cell phenotype and function (a composite measure of (I) NK cell frequency and (II) expression of activation and inhibitory markers (III) IFN-y production upon IL-12/IL-18 stimulation and (IV) Perforin granzyme production | 1 year

SECONDARY OUTCOMES:
Gene expression levels of the type I IFN signaling pathway on whole blood samples measured by multiplex | 1 year
Gene expression levels of leukocyte populations before, during and after treatment measured by microarray | 2 years
Serum cytokines levels using multiplex platforms LUMINEX -100 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rob de Knegt, M.D., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Derived] Spaan M, van Oord G, Kreefft K, Hou J, Hansen BE, Janssen HL, de Knegt RJ, Boonstra A. Immunological Analysis During Interferon-Free Therapy for Chronic Hepatitis C Virus Infection Reveals Modulation of the Natural Killer Cell Compartment. J Infect Dis. 2016 Jan 15;213(2):216-23. doi: 10.1093/infdis/jiv391. Epub 2015 Jul 28. PMID 26223768